CLINICAL TRIAL: NCT05320848
Title: Value of Cardiac Rehabilitation on the Treatment of Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SY-CSF-001
Record Dates: First submitted 2021-08-04; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Rehabilitation
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): the patients treated with cardiac rehabilitation intervention.
  Interventions: Behavioral: cardiac rehabilitation
- Control group (No Intervention): the patients treated without cardiac rehabilitation intervention.

INTERVENTIONS:
Behavioral: cardiac rehabilitation — Cardiac rehabilitation is a valuable treatment for patients with a broad spectrum of cardiac disease.
  Arms: Treatment group

SUMMARY:
Cardiac rehabilitation is a valuable treatment for patients with a broad spectrum of cardiac disease. Current guidelines support its use in patients after acute coronary syndrome, coronary artery bypass grafting, coronary stent placement, valve surgery, and stable chronic systolic heart failure. Its use in these conditions is supported by a robust body of research demonstrating improved clinical outcomes. Despite this evidence, cardiac rehabilitation referral and attendance remains low and interventions to increase its use need to be developed.

DETAILED DESCRIPTION:
The trial was conducted in Shenzhen in China. This study will recruit 100 patients with cardiovascular disease with a median and minimum follow-up of 24 and 6 months. Patients will be individually randomized to receive either a cardiac rehabilitation program (n = 50) or enhanced standard care involving educational advice (n = 50). The co-primary outcomes are: 1) first occurrence of major adverse cardiovascular events (MACE) (composite of all-cause mortality, myocardial infarction, stroke, or emergency cardiovascular hospitalization); and 2) self-rated health on the Quality of Life-5 Dimensions-5 Level visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease

Exclusion Criteria:

* Incalculable TFC
* Coronary artery spasm or ectasia
* LV ejection fraction < 52% in males or < 54% in females
* Abnormal heart structure (congenital heart disease, cardiomyopathies, or valvular dysfunction)
* Pericardial disease (pericardial effusion or constrictive pericarditis)
* Previous history of myocardial infarction
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 105 mmHg)
* Hyperthyroidism
* Hypothyroidism
* Malignancy
* Autoimmune disease
* Infection
* Pulmonary, hepatic, and renal disorders
* Haematological disorders (anaemia, bone marrow involved by neoplastic disease, or red blood cell transfusions)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
first occurrence of major adverse cardiovascular events (MACE) | 3 years
  first occurrence of major adverse cardiovascular events (MACE) (composite of all-cause mortality, myocardial infarction, stroke, or emergency cardiovascular hospitalization)
maximum oxygen uptake | 3 years
  maximum oxygen uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson L, Thompson DR, Oldridge N, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2016 Jan 5;2016(1):CD001800. doi: 10.1002/14651858.CD001800.pub3. PMID 26730878
- [Background] Ruano-Ravina A, Pena-Gil C, Abu-Assi E, Raposeiras S, van 't Hof A, Meindersma E, Bossano Prescott EI, Gonzalez-Juanatey JR. Participation and adherence to cardiac rehabilitation programs. A systematic review. Int J Cardiol. 2016 Nov 15;223:436-443. doi: 10.1016/j.ijcard.2016.08.120. Epub 2016 Aug 13. PMID 27557484
- [Background] Wong WP, Feng J, Pwee KH, Lim J. A systematic review of economic evaluations of cardiac rehabilitation. BMC Health Serv Res. 2012 Aug 8;12:243. doi: 10.1186/1472-6963-12-243. PMID 22873828
- [Background] Ragupathi L, Stribling J, Yakunina Y, Fuster V, McLaughlin MA, Vedanthan R. Availability, Use, and Barriers to Cardiac Rehabilitation in LMIC. Glob Heart. 2017 Dec;12(4):323-334.e10. doi: 10.1016/j.gheart.2016.09.004. Epub 2017 Mar 13. PMID 28302548
- [Background] Edwards K, Jones N, Newton J, Foster C, Judge A, Jackson K, Arden NK, Pinedo-Villanueva R. The cost-effectiveness of exercise-based cardiac rehabilitation: a systematic review of the characteristics and methodological quality of published literature. Health Econ Rev. 2017 Oct 19;7(1):37. doi: 10.1186/s13561-017-0173-3. PMID 29052044